CLINICAL TRIAL: NCT00419042
Title: A Multicenter Randomized Phase II Trial in NSCLC Stage IV et IIIB in Elderly Dependent Patients With Evaluation of the Sequence Gemcitabine First Line Followed by Erlotinib When Progression Versus Erlotinib First Line Followed by Gemcitabine When Progression.
Brief Title: Elderly Dependent Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Groupe Francais De Pneumo-Cancerologie (Other)
Responsible Party: Sponsor
Other Study IDs: GFPC 05-05
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2010-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: cancer; Lung cancer; None small-cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Lung Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: TARCEVA — Tarceva (150 mg) is a pill you take once a day -- every day -- to help treat non-small cell lung cancer.
  Other Names: Erlotinib
Drug: Gemzar — GEMZAR by mixing it into a solution and giving it through a needle into a vein-called intravenous infusion (IV). This will take about 30 minutes
  Other Names: Gemcitabine

SUMMARY:
The purpose of this study is in non small-cell lung cancer stage IV et IIIB (T4 with pleural effusion) in elderly dependent patients with evaluation of the sequence Gemcitabine first line followed by Erlotinib when progression versus Erlotinib first line followed by Gemcitabine when progression

DETAILED DESCRIPTION:
A multicenter phase II trial,prospective,randomized,open,non comparative

ELIGIBILITY:
Inclusion Criteria:

* Age > 65
* Comorbidities score, PS and frailty score according to table 1
* No dementia, faecal or urinary incontinence, repeated falls
* ADL = 0, IADL = 0-1
* Life expectancy at least 12 weeks
* Creatinin clearance > = 30 ml/mn (according to Cockcrofts-Gault formula)
* Competency to give written informed consent
* Haematological functions as follows : neutrophiles count > 1.5 x 109/l and platelets > 100 x 109/l hemoglobin > 9,5 g/dl - Hepatic function as follows : Bilirubin < 1,25 LNS ASAT / ALAT <5 x NAlcPh <5 x N
* PS < 3
* cerebral metastasis eligible if asymptomatic
* Histologically or cytologically confirmed NSCLC
* Stage IV/IIIB4 (T4 with pleural effusion)
* No prior chemotherapy
* relapses of previous NSCLC treated by surgery or radiotherapy are eligible, if the target is measurable out of initial radiotherapy field and if cytological or histological proof
* At least one measurable target lesion by RECIST guidelines

Exclusion Criteria:

* symptomatic cerebral metastasis
* Any severe comorbidity calculated by Charlson score according to table 1
* ADL > 0 and IADL > 1- performance status >2 (ECOG)
* peripheral neuropathy grade 2 or more
* dementia, repeated falls, urinary or faecal incontinence
* contra-indication to corticosteroids
* contra indication to a product of this study
* unwilling or unable to comply with study requirements, for personal, family, sociologic, geographic or any other reason
* inability of the subject to give written informed consent
* lack of liberty following legal or administrative decision
* hypersensitivity to polysorbate
* hypersensitivity to erlotinib or any excipients of this product
* unusual hereditary disorders, as galactosemia, deficit in lactase and syndrome of malabsorption in glucose or galactose
* participation in concomitant clinical trial
* bronchioloalveolar or neuroendocrine or composite carcinoma
* superior vena cava syndrome

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with non small-cell lung cancer stage IV et IIIB (T4 with pleural effusion) in elderly dependent patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-07; Primary Completion 2006-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé LECAER, Doctor, Principal Investigator — Groupe Francais De Pneumo-Cancerologie
Locations (23):
- France (23):
  - Site 12, Aix-en-Provence
  - Site 05, Bastia
  - Site 22, Beauvais
  - Site 43, Caen
  - Site 30, Charleville-Mézières
  - Site 33, Créteil
  - Site 07, Draguignan
  - Site 32, Elbeuf
  - Site 04, Gap
  - Site 41, Le Chesnay
  - Site 00, Limoges
  - Site 25, Mantes-la-Jolie
  - Site 06, Marseille
  - Site 27, Martigues
  - Site 01, Meaux
  - Site 42, Orléans
  - Site 26, Paris
  - Site 19, Périgueux
  - Site 02, Reims
  - Site 20, Rennes
  - Site 17, Rouen
  - Site 14, Toulon
  - Site 11, Villefranche-sur-Saône

REFERENCES:
- See also: Groupement Francais de Pneumo-cancérologie — http://www.g-f-p-c.org